CLINICAL TRIAL: NCT04939688
Title: Concordance Between Ultra-low Dose (ULD) and Conventional Standard Dose CT Scans in the Search for Traumatic Brain Injury at the Emergency Department
Brief Title: Concordance Between Ultra-low Dose (ULD) and Standard Dose CT Scans in the Search for Traumatic Brain Injury
Acronym: ULD-CRANE
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Recruitment difficulties
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: NIMAO/2020-1/NM-01
Record Dates: First submitted 2021-06-17; First posted 2021-06-25 (Actual); Last update posted 2025-03-10 (Actual); Status verified 2025-03

CONDITIONS: Head Injuries, Penetrating; Head Injuries, Closed
MeSH Terms: conditions — Head Injuries, Penetrating; Head Injuries, Closed

STUDY DESIGN:
Intervention Model Description: All patients requiring investigation of traumatic injuries after moderate or severe head trauma as identified at the emergency department. All patients will receive a standard dose CT scan of the skull according to the usual management, as well as a ULD scan of the same area, performed specifically for the needs of the study, following a pre-established standardized protocol. The center's radiologist will interpret the conventional CT scan in real time for patient diagnosis and management, but this interpretation will not be used in the study. The patient will then be redirected to the emergency department for his or her usual management.
Masking Description: All patients will have the benefit of two CT scans : one normal dose and one ultra low-dose. However, the results of scans will be interpreted by two independent radiologists (senior and junior) who do not know whether the scan has been done with the normal, classic dose or with the ultra low-dose protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients requiring a CT scan in the search for cranial lesions following head trauma (Experimental): All patients will undergo both conventional dose AND ultra low-dose CT scans in the search for cranial lesions following head trauma.
  Interventions: Radiation: Conventional dose AND ultra low-dose CT scanning in the search for cranial lesions

INTERVENTIONS:
Radiation: Conventional dose AND ultra low-dose CT scanning in the search for cranial lesions — As well as undergoing the usual, conventional radiation dose CT scan, these patients will also undergo ultra low-dose CT scanning in the search for cranial lesions.

SUMMARY:
The aim of this research is to evaluate the diagnostic concordance of ultra low-dose and standard dose reconstructed computed tomography acquisitions using the ADMIRE algorithm to search for intracranial lesions - both hemorrhagic and bone lesions - in trauma patients at the emergency department. The study will also evaluate the diagnostic performance of the two protocols, as well as the speed of image reading. For the first time, acquisitions ≤ 10 mGy (lower value than reported in the literature) will be performed with top-of-the-range scanners available in the emergency room to search for intracranial lesions. These scanners are equipped with the latest generation of ADMIRE iterative algorithms.

DETAILED DESCRIPTION:
Head trauma is a common reason for consultation at the casualty department. The CT computed tomography scan is the standard examination leading to rapid patient management (admission to intensive care or neurosurgical management). The prevalence of traumatic lesions, intracranial bleeding or fractures, is estimated at 90% in moderate or severe head trauma patients, justifying the systematic use of a CT scan.

X-ray exposure from CT scanners is among the highest (order of May 23, 2019 for the Diagnostic Reference Levels, DRL). Radiation protection principles therefore require continuous optimization of acquisition procedures to ensure the lowest possible dose to the patient whilst maintaining satisfactory image quality for diagnosis. In recent years, technological innovations have been developed to optimize the dose delivered to the scanner, such as iterative reconstructions. Numerous studies on image quality and anthropomorphic phantoms and on cadavers have been performed at the imaging department of Nîmes University Hospital. Subsequently, feasibility studies have been conducted on patients, highlighting the use of the ultra low-dose scanner to detect common pathologies. These studies have made it possible to set up "ultra-low dose" acquisitions for several pathologies with an effective dose level close to a standard radiographic examination. These ultra low-dose acquisitions are now routinely used in our clinical practice for thoracic, spine, pelvis and proximal femurs, extremities and abdomino-pelvic explorations.

In the literature, some studies have explored the feasibility of ultra low-dose acquisitions for ear, nose and throat or skull explorations. Our study is in the context of evaluating ULD acquisitions for skull CT for traumatic intracranial lesions. The study by Corcuera-Solano et al. (2014) showed the feasibility of ULD acquisitions (Scanographic Dose Index in Volume, mean SDVI = 15.5 mGy) compared to standard acquisition (mean SDVI = 48.38 mGy) in the follow-up of a heterogeneous group of patients admitted to the neurosurgical intensive care unit, without evaluating the diagnostic performance of the two acquisitions. In this study, the Siemens scanner used was equipped with a 2nd generation iterative reconstruction algorithm (SAFIRE).

A 3rd generation algorithm has since been developed (ADMIRE) allowing an improvement in image texture, thus favoring the use of ultra low-dose acquisition for structures with lower spontaneous contrast such as the encephalon. We believe it would therefore be possible to search for intracranial lesions in trauma patients using ultra low-dose protocols, which should make it possible to reduce the doses delivered to the patient whilst maintaining sufficient image quality for diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* All patients in an emergency situation with a head trauma requiring a scan, i.e. moderate or severe skull trauma, Group 1 or 2 according to the Brain Trauma Task Force classification (Guidelines for management of severe head injury. J Neurotrauma 2000 ; 17 : 507-11) as described by P. Schoettker et al. 2001).
* Patient with an isolated skull trauma or polytraumatized patient including skull trauma.
* Patient capable of giving informed consent or for whom a person of confidence or legal representative / family member has given informed consent and signed the consent form on the patient's behalf if the patient has been included in an emergency.
* Patients affiliated to or beneficiary of a health insurance scheme.
* All adult patients aged 18 or over.

Exclusion Criteria:

* Patients already taking part in another study for which it is not allowed to participate in other clinical studies.
* Patients in an exclusion period determined by another study.
* Patients who are pregnant, breastfeeding or about to give birth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-26 (Actual); Primary Completion 2021-07-19 (Actual); Study Completion 2021-07-19 (Actual)

PRIMARY OUTCOMES:
Presence of at least one extradural hematoma found on the standard dose CT-scan | Day 0
  YES/NO
Presence of at least one extradural hematoma found on the ultra low-dose CT-scan | Day 0
  YES/NO
Presence of at least one subarachnoid hemorrhage found on the standard dose CT-scan | Day 0
  YES/NO
Presence of at least one subarachnoid hemorrhage found on the ultra low-dose CT-scan | Day 0
  YES/NO
Presence of at least one subdural hematoma found on the standard dose CT-scan | Day 0
  YES/NO
Presence of at least one subdural hematoma found on the ultra low-dose CT-scan | Day 0
  YES/NO
Presence of at least one intraparenchymal hemorrhage found on the standard dose CT-scan | Day 0
  YES/NO
Presence of at least one intraparenchymal hemorrhage found on the ultra low-dose CT-scan | Day 0
  YES/NO

SECONDARY OUTCOMES:
A. Presence of at least one bone lesion in the skull, arch or face found on the standard dose CT-scan | Day 0
  YES/NO
A. Presence of at least one bone lesion in the skull, arch or face found on the ultra low-dose CT-scan | Day 0
  YES/NO
B. Presence of at least one intracranial hemorrhagic lesion found on the standard dose CT-scan | Day 0
  YES/NO
B. Presence of at least one intracranial hemorrhagic lesion found on the ultra low-dose CT-scan | Day 0
  YES/NO
C. Presence of at least one cranial bone lesion found on the standard dose CT-scan | Day 0
  YES/NO
C. Presence of at least one cranial bone lesion found on the ultra low-dose CT-scan | Day 0
  YES/NO
D. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion found on the standard dose CT-scan according to the radiologist. | Day 0
  YES/NO
D. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion found on the ultra low-dose CT-scan according to the radiologist. | Day 0
  YES/NO
E. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion found on the standard dose CT-scan | Day 0
  YES/NO
E. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion found on the ultra low-dose CT-scan | Day 0
  YES/NO
Fi.Radiologist's appreciation of the standard dose CT-scan: image quality | Day 0
  A scale of 1 - 4 will be used (1 = interpretable, 2 = interpretable despite a slight technical problem (centering, movement, constants) 3 = completely interpretable despite a slight technical problem, 4 = no technical problems)
Fi.Radiologist's appreciation of the ultra low-dose CT-scan: image quality | Day 0
  A scale of 1 - 4 will be used (1 = interpretable, 2 = interpretable despite a slight technical problem (centering, movement, constants) 3 = completely interpretable despite a slight technical problem, 4 = no technical problems)
Fii.Radiologist's appreciation of the standard dose CT-scan: diagnostic quality | Day 0
  A scale of 1 - 5 will be used (1 = unacceptable, 2 = sub-optimal, 3 = acceptable, 4 = above average, 5 = excellent)
Fii.Radiologist's appreciation of the ultra low-dose CT-scan: diagnostic quality | Day 0
  A scale of 1 - 5 will be used A scale of 1 - 5 will be used (1 = unacceptable, 2 = sub-optimal, 3 = acceptable, 4 = above average, 5 = excellent)
Fiii.Radiologist's appreciation of the standard dose CT-scan: level of confidence | Day 0
  A scale of 1 - 5 will be used (1 = very poor, 2 = poor, 3 = moderate, 4 = high, 5 = excellent)
Fiii.Radiologist's appreciation of the ultra low-dose CT-scan: level of confidence | Day 0
  A scale of 1 - 5 will be used (1 = very poor, 2 = poor, 3 = moderate, 4 = high, 5 = excellent)
G. Total dose of X-rays delivered with the standard dose CT-scan : DLP | Day 0
  DACS (Dose Archiving and Communication System) will be used to measure Dose Length Product (DLP) measured in mGy*cm
G. Total dose of X-rays delivered with the ultra low-dose CT-scan : DLP | Day 0
  DACS (Dose Archiving and Communication System) will be used to measure Dose Length Product (DLP) measured in mGy*cm
G. Total dose of X-rays delivered with the standard dose CT-scan : CTDI | Day 0
  DACS (Dose Archiving and Communication System) will be used to measure Computed Tomography Dose Index in mGy
G. Total dose of X-rays delivered with the ultra low-dose CT-scan : CTDI | Day 0
  DACS (Dose Archiving and Communication System) will be used to measure Computed Tomography Dose Index in mGy
H. Interpretation time with the standard dose CT-scan | Day 0
  The time taken to interpret the images will be measured in minutes
H. Interpretation time with the ultra low-dose CT-scan | Day 0
  The time taken to interpret the images will be measured in minutes
I. Performance of standard dose CT-scan for polytrauma patients. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion. | Day 0
  YES/NO
I. Performance of the ultra low-dose CT-scan for patients with skull trauma alone. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion | Day 0
  YES/NO
I. General performance of the ultra low-dose CT-scan for polytrauma patients: Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion | Day 0
  YES/NO
I. General performance of the standard dose CT-scan for patients with skull trauma alone. Presence of at least one intracranial hemorrhagic lesion and presence of at least one bone lesion | Day 0
  YES/NO

OTHER OUTCOMES:
Patient's age | Day 0
  In years
Patient's weight | Day 0
  In kilos
Patient's height | Day 0
  In cm
Patient's Body Mass Index | Day 0
  The patient's Body Mass Index will be calculated by computer according to the patient's weight and height (in Kg/m²)
Type of trauma | Day 0
  The type of trauma will be recorded
Circumstances of trauma | Day 0
  The circumstances of the trauma will be recorded

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas MENJEOT DE CHAMPFLEUR, Principal Investigator — Nîmes University Hospital
Locations (1):
- Nîmes University Hospital, Nîmes, Gard, France

REFERENCES:
- [Background] Greffier J, Fernandez A, Macri F, Freitag C, Metge L, Beregi JP. Which dose for what image? Iterative reconstruction for CT scan. Diagn Interv Imaging. 2013 Nov;94(11):1117-21. doi: 10.1016/j.diii.2013.03.008. Epub 2013 Jun 22. PMID 23796396
- [Background] Greffier J, Macri F, Larbi A, Fernandez A, Khasanova E, Pereira F, Mekkaoui C, Beregi JP. Dose reduction with iterative reconstruction: Optimization of CT protocols in clinical practice. Diagn Interv Imaging. 2015 May;96(5):477-86. doi: 10.1016/j.diii.2015.02.007. Epub 2015 Mar 19. PMID 25797211
- [Background] Larbi A, Orliac C, Frandon J, Pereira F, Ruyer A, Goupil J, Macri F, Beregi JP, Greffier J. Detection and characterization of focal liver lesions with ultra-low dose computed tomography in neoplastic patients. Diagn Interv Imaging. 2018 May;99(5):311-320. doi: 10.1016/j.diii.2017.11.003. Epub 2018 Feb 1. PMID 29396085
- [Background] Maas AI, Hukkelhoven CW, Marshall LF, Steyerberg EW. Prediction of outcome in traumatic brain injury with computed tomographic characteristics: a comparison between the computed tomographic classification and combinations of computed tomographic predictors. Neurosurgery. 2005 Dec;57(6):1173-82; discussion 1173-82. doi: 10.1227/01.neu.0000186013.63046.6b. PMID 16331165
- [Background] Macri F, Greffier J, Pereira F, Rosa AC, Khasanova E, Claret PG, Larbi A, Gualdi G, Beregi JP. Value of ultra-low-dose chest CT with iterative reconstruction for selected emergency room patients with acute dyspnea. Eur J Radiol. 2016 Sep;85(9):1637-44. doi: 10.1016/j.ejrad.2016.06.024. Epub 2016 Jul 1. PMID 27501900
- [Background] Macri F, Greffier J, Pereira FR, Mandoul C, Khasanova E, Gualdi G, Beregi JP. Ultra-low-dose chest CT with iterative reconstruction does not alter anatomical image quality. Diagn Interv Imaging. 2016 Nov;97(11):1131-1140. doi: 10.1016/j.diii.2016.06.009. Epub 2016 Jul 20. PMID 27451261
- [Background] Widmann G, Juranek D, Waldenberger F, Schullian P, Dennhardt A, Hoermann R, Steurer M, Gassner EM, Puelacher W. Influence of Ultra-Low-Dose and Iterative Reconstructions on the Visualization of Orbital Soft Tissues on Maxillofacial CT. AJNR Am J Neuroradiol. 2017 Aug;38(8):1630-1635. doi: 10.3174/ajnr.A5239. Epub 2017 Jun 8. PMID 28596194